CLINICAL TRIAL: NCT03908580
Title: A Prospective, Multi-center, Single Arm, Open-label, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of MEDITOXIN® in Treatment of Post Stroke Upper Limb Spasticity
Brief Title: MEDITOXIN® Treatment in Subjects With Post-Stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT_PRT_ST02
Record Dates: First submitted 2019-03-26; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Spasticity, Muscle
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditoxin® (Experimental): Botulinum toxin type A was intramuscularly injected up to 360U and up to 4 sites, depending on the muscle size.
  Interventions: Drug: Meditoxin

INTERVENTIONS:
Drug: Meditoxin — Meditoxin® (Botulinum toxin type A) was injected up to 360 U.
  Other Names: Neuronox®

SUMMARY:
This study is "A Prospective, Multi-center, Single Arm, Open-label, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of MEDITOXIN® in Treatment of Post Stroke Upper Limb Spasticity".

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 20 years.
2. Subjects that was diagnosed with stroke at least 1 month before participating in the clinical trial.
3. Subjects with MAS score of ≥2 for local muscle spasticity of wrist flexor.

Exclusion Criteria:

1. Subjects with generalized neuromuscular junction disorder (ex: myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, etc.).
2. Subjects with fixed joint, muscle contracture, or atrophy in the treatment area.
3. Subjects with botulinum toxin treatment within 3 months before administration of the investigational product.
4. Known immunization or hypersensitivity to any botulinum toxin preparations.
5. Subjects who have recieved the following treatments within 4 weeks from screening: Muscle relaxants, Benzodiazepines, Aminoglycosides, Other antibiotics, Anticholinergics

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09-06 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Change in muscle tone determined by MAS (Modified Ashworth Scale) of wrist flexor | 4 weeks
  Change in muscle tone determined by MAS (Modified Ashworth Scale: Measures resistance during passive soft-tissue stretching; score 0 to 4, 4 being most difficult passive movement) of wrist flexor in subjects with post stroke upper limb spasticity at week 4 after administration compared to baseline.

SECONDARY OUTCOMES:
Change in muscle tone determined by MAS (Modified Ashworth Scale) of elbow flexor and finger flexor | 4 weeks, 16 weeks, and 4 weeks after re-visit
  Change in muscle tone determined by MAS (Modified Ashworth Scale: Measures resistance during passive soft-tissue stretching; score 0 to 4, 4 being most difficult passive movement) of elbow flexor and finger flexor at week 4 and 16 after administration compared to baseline, and at 4 weeks after re-administration compared to the time of re-visit.
Change in muscle tone determined by MAS (Modified Ashworth Scale) of wrist flexor | 16 weeks, and 4 weeks after re-visit
  Change in muscle tone determined by MAS (Modified Ashworth Scale: Measures resistance during passive soft-tissue stretching; score 0 to 4, 4 being most difficult passive movement) of wrist flexor at week 16 after administration compared to baseline, and at 4 weeks after re-administration compared to the time of re-visit.
The effective rate of wrist flexor, elbow flexor, and finger flexor | 4 weeks, 16 weeks, and 4 weeks after re-visit
  The effective rate of wrist flexor, elbow flexor, and finger flexor at week 4 and 16 compared to baseline and at week 4 after re-administration compared to re-visit, defining the muscle with MAS (Modified Ashworth Scale: Measures resistance during passive soft-tissue stretching; score 0 to 4, 4 being most difficult passive movement) score of ≥1 among the wrist flexor, elbow flexor, and finger flexor muscles as responders when the MAS is reduced by 1 score compared to baseline (week 0).
Change in DAS (Disability Assessment Scale) score | 4 weeks, 16 weeks, and 4 weeks after re-visit
  Change in score of goal assessment section in DAS (Disability Assessment Scale: Measures disability associated with upper limb spasticity in patients; score 0 to 3, 3 being the most severe disability) at week 4 and 16 compared to baseline and at week 4 after re-administration compared to re-visit.
Change in QOL (SF-36v2; Quality of Life) score | 4 weeks, 16 weeks, and 4 weeks after re-visit
  Change in score of Short Form 36 ver.2 (SF-36v2; Quality of Life, QOL: a questionnaire with 36 questions regarding general health change affecting patient's quality of life; score from 1 up to 5, from minimum to high impact on quality of life) at week 4 and 16 compared to baseline and at week 4 after re-administration compared to re-visit.
Subject's or caregiver's global assessment | 4 weeks, 16 weeks, and 4 weeks after re-visit
  Subject's or caregiver's global assessment (rating from -3 to +3 on the overall treatment effect, with +3 being very satisfied with treatment) at week 4 and 16 compared to baseline and at week 4 after re-administration compared to re-visit.
Number of participants with Adverse Events (AEs) to assess safety of investigational product. | Through study completion, an average of 1 year
  Safety of IP assessed by the number of partiicipants with adverse events determined by MedDra ver 16.0 from enrollment to the end of study.